CLINICAL TRIAL: NCT04201743
Title: A Prospective, Double-Blinded, Randomized Controlled Trial of an Amniotic Membrane Injection Comparing Two Doses (1 mL and 2mL Injection) in the Treatment of Osteoarthritis of the Knee
Brief Title: An Amniotic Membrane Injection Comparing Two Doses (1 mL and 2mL Injection) in the Treatment of Osteoarthritis of the Knee
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Resources limited secondary to COVID-19 pandemic.
Sponsor: Illinois Center for Orthopaedic Research and Education (Other)
Responsible Party: Principal Investigator, Ronak M. Patel, President, Illinois Center for Orthopaedic Research and Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 199608
Record Dates: First submitted 2019-12-08; First posted 2019-12-17 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Amniotic membrane; Allograft
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Data will be prospectively collected on all injectable acellular amniotic membrane derived allograft knee performed at our institute.
  Inclusion criteria will be all patients age between 21 and 80 years with a diagnosis of osteoarthritis (OA) defined as Grade 1 to 3 on the Kellgren Lawrence grading scale.
  Methods for collecting data will be through validated patient-reported outcome tools that the patient will complete pre-injection and at specified time intervals after injection: 90 days, 180 days and 365 days.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 mL NyDYN injection (Active Comparator): 30 patients (out of 60) will be doubled blinded randomized to this arm and get 1 mL NyDYN injection.
  Interventions: Drug: Acellular amniotic membrane derived allograft injection (NuDYN)
- 2 mL NyDYN injection (Active Comparator): 30 patients (out of 60) will be doubled blinded randomized to this arm and get 2 mL NyDYN injection.
  Interventions: Drug: Acellular amniotic membrane derived allograft injection (NuDYN)

INTERVENTIONS:
Drug: Acellular amniotic membrane derived allograft injection (NuDYN) — Injectable acellular amniotic membrane derived allograft (NuDYN) through routine follow-up with physical examination, pain, function and quality of life measurements and compare dose effects (1 mL versus 2 mL of NuDYN injection) in the treatment of knee osteoarthritis.

SUMMARY:
The purpose of this study is to determine the dose effect of a single injectable acellular amniotic membrane derived allograft injection for the treatment of knee osteoarthritis and to confirm whether the use of 2 mL of the same amniotic injection offers a statistically significant advantage over the 1 mL injection.

DETAILED DESCRIPTION:
It is a prospective, double blinded, Randomized Controlled Trial study. Data will be prospectively collected of all injectable acellular amniotic membrane derived allograft knee performed at our institute (1 vs 2 mL).

60 subjects will be enrolled in this study. Subjects will be randomized 1:1 in treatment arms.

Each of the patient will be treated with one time injection to the knee. Methods for collecting data will be through validated patient-reported outcome tools (KOOS, VAS and WOMAC questionnaire) that the patient will complete pre-injection and at specified time intervals after injection: 90 days, 180 days and 365 days.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 to 80 years
* Diagnosis of osteoarthritis (OA) defined as Grade 1 to 3 on the Kellgren Lawrence grading scale

Exclusion Criteria:

* Subject has a diagnosis of osteoarthritis (OA) defined as Grade 4 on the Kellgren Lawrence grading scale
* BMI greater than 40 kg/m2
* Subject has active infection at the injection site
* Symptomatic OA of the contralateral knee or of either hip that is not responsive to acetaminophen (Tylenol) and requires other therapy.
* Subject has rheumatoid arthritis, psoriatic arthritis or has been diagnosed with any other disorder that is the primary source of their knee pain, including but not limited to: osteonecrosis, radiculopathy, bursitis, tendinitis, tumor or cancer
* Subject has documented history of gout or pseudo-gout
* Subject has an autoimmune disease or known history of having Acquired Immunodeficiency Syndromes (AIDS) or HIV
* Subject has received any of the following to the target knee:

  1. Intra-articular hyaluronic acid (HA) injection within 12 weeks prior to screening
  2. Intra-articular cortisone (steroid/corticosteroid) injection into the knee joint within 12 weeks of treatment
  3. Steroid or platelet rich plasma (PRP) injection within 12 weeks prior to screening
  4. Has had or is planning to have major surgery or arthroscopy in the target knee within 26 weeks of treatment
* History of partial or total knee arthroplasty
* Subject has used an investigational drug, device or biologic within 12 weeks prior to treatment
* Subject has a history of immunosuppressive or chemotherapy in the last 5 years
* Subject has had prior radiation at the site
* Subject is currently taking narcotic medication for any reason.
* Subject is pregnant or plans to become pregnant within 365 days of treatment
* Subject has any significant medical condition that, in the opinion of the Investigator, would interfere with protocol evaluation and participation
* Subject is a worker's compensation patient
* Subject is a prisoner

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoints using Validated patient-reported outcome tools questionnaires | 180 days
  Knee injury and Osteoarthritis Outcome Score (KOOS)- assess five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. It is a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Primary Efficacy Endpoints using Validated patient-reported outcome tools questionnaires | 180 days
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)- assess the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. it is a 0 (worst)-96 scale (best).
Primary Efficacy Endpoints using Validated patient-reported outcome tools questionnaires | 180 days
  Visual Analogue Scale (VAS)- assess pain, It is a 0-100 scale. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Exploratory Endpoint using Validated patient-reported outcome tools questionnaires | 90, 180 and 365 days
  Change from baseline Knee injury and Osteoarthritis Outcome Score (KOOS)- assess five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. It is a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Exploratory Endpoint using Validated patient-reported outcome tools questionnaires | 90, 180 and 365 days
  Change from baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)- assess the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. it is a 0 (worst)-96 scale (best).
Exploratory Endpoint using Validated patient-reported outcome tools questionnaires | 90, 180 and 365 days
  Change from baseline Visual Analogue Scale (VAS)- assess pain, It is a 0-100 scale. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Patel, MD, Principal Investigator — Illinois Center for Orthopedic Research and Education (iCORE)
Locations (1):
- Hinsdale Orthopaedic Associates, Westmont, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riboh JC, Saltzman BM, Yanke AB, Cole BJ. Human Amniotic Membrane-Derived Products in Sports Medicine: Basic Science, Early Results, and Potential Clinical Applications. Am J Sports Med. 2016 Sep;44(9):2425-34. doi: 10.1177/0363546515612750. Epub 2015 Nov 19. PMID 26585668
- [Background] Vines JB, Aliprantis AO, Gomoll AH, Farr J. Cryopreserved Amniotic Suspension for the Treatment of Knee Osteoarthritis. J Knee Surg. 2016 Aug;29(6):443-50. doi: 10.1055/s-0035-1569481. Epub 2015 Dec 18. PMID 26683979